CLINICAL TRIAL: NCT01512888
Title: A Pilot Feasibility Study of Gene Transfer for X-Linked Severe Combined Immunodeficiency in Newly Diagnosed Infants Using a Self-Inactivating Lentiviral Vector to Transduce Autologous CD34+ Hematopoietic Cells
Brief Title: Gene Transfer for X-Linked Severe Combined Immunodeficiency in Newly Diagnosed Infants
Acronym: LVXSCID-ND
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: voluntary hold
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Assisi Foundation (Other); California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LVXSCID-ND; P01HL053749 (NIH)
Record Dates: First submitted 2012-01-13; First posted 2012-01-19 (Estimated); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Severe Combined Immunodeficiency Disease, X-linked
Keywords: SCID; SCID-X1; X-linked SCID; immunodeficiency; gene therapy
MeSH Terms: conditions — X-Linked Combined Immunodeficiency Diseases; Immunologic Deficiency Syndromes | interventions — Busulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Treatment (Experimental): Participants will undergo a bone marrow harvest in the operating room to obtain bone marrow cells. Cells will be isolated and purified utilizing the CliniMacs device. These cells will undergo vector transduction with the lentiviral vector that contains a normal copy of the γc gene gene (CL20-i4-EF1α-hγc-OPT) and then the transduced cells will be reinfused back into the patient. Participants will receive a conditioning regimen of busulfan 3 days prior and 2 days prior to infusion of vector-corrected cells.intervention: CL20-i4-EF1α-hγc-OPT
  Interventions: Genetic: CL20-i4-EF1α-hγc-OPT; Drug: Busulfan; Device: CliniMacs

INTERVENTIONS:
Genetic: CL20-i4-EF1α-hγc-OPT — Participants will undergo infusion with autologous CD34+ bone marrow cells transduced with a lentiviral vector that contains a normal copy of the human γc gene.
  Other Names: self inactivating lentiviral vector; IND 14570
Drug: Busulfan — Given intravenously (IV).
  Other Names: Busulfex®; Myleran®
Device: CliniMacs — Isolation and purification of CD34+ stem cells will be done after the unmodified frozen backup is obtained and in accordance with our FDA IND and in accordance with the CliniMacs manual of operations.

SUMMARY:
SCID-X1 is a genetic disorder of blood cells caused by DNA changes in a gene that is required for the normal development of the human immune system. The purpose of this study is to determine if a new method, called lentiviral gene transfer, can be used to treat SCID-X1. This method involves transferring a normal copy of the common gamma chain gene into the participant's bone marrow stem cells. The investigators want to determine if the procedure is safe, whether it can be done according to the methods they have developed, and whether the procedure will provide a normal immune system for the patient. It is hoped that this type of gene transfer may offer a new way to treat children with SCID-X1 that do not have a brother or sister who can be used as a donor for stem cell transplantation.

DETAILED DESCRIPTION:
Bone marrow CD34+ cells will be obtained in the operating room, transduced with the lentiviral vector that contains a normal copy of the γc gene, and reinfused without any myeloreductive conditioning. Participants will be monitored for hematopoietic recovery from busulfan and for severe adverse events for 42 days post gene therapy. The primary endpoint assessing the efficacy of this approach will be T-cell immune reconstitution 52 weeks (± 4) weeks after transplantation. Continued and detailed evaluation of all aspects of immune reconstitution, protocol-related toxicity, and retroviral integration sites will also be performed. This study will evaluate the first use of a SIN lentiviral vector for the treatment of SCID-X1 and may lead to a new form of therapy that could be applied to the majority of newly diagnosed patients.

OBJECTIVES

Assess the safety, feasibility and efficacy of lentiviral gene transfer in newly diagnosed SCID-X1 patients transplanted with autologous CD34+ cells that have been transduced with a self-inactivating lentiviral vector (CL20-i4-EF1α-hγc-OPT) expressing a γc gene.

Primary Objective 1: Evaluate the safety and feasibility of infusing at least 1 million transduced CD34+ cells per kilogram of body weight in SCID-X1 infants.

Primary Objective 2: Evaluate the efficacy of lentiviral gene transfer for inducing significant T-cell reconstitution 52 weeks (± 4 weeks) after transplantation. Significant reconstitution of T cells is defined as at least 2 of the following 3 criteria being present:

* The development of T-cell proliferative responses to phytohemagglutinin (PHA) that are ≥ 50% the value seen in normal controls
* ≥ 1000 autologous CD3+ T-cells/μl in the peripheral blood
* ≥ 500 autologous CD4+ T-cells/μl in the peripheral blood
* ≥ 200 autologous CD4+ CD45RA T-cells/μl in the peripheral blood

OTHER PRE-SPECIFIED OBJECTIVES:

* Correlate busulfan and its metabolite pharmacokinetics with toxicity, efficacy, engraftment of vector-transduced cells, and event-free survival and overall survival.
* Evaluate the efficacy of busulfan dose-targeting with busulfan administration every 24 hours for a total of 2 doses in order to achieve a cumulative busulfan area under the curve of 22 mg*hr/L.
* Evaluate B-cell function during longterm follow-up of protocol patients. Evaluation will include γc expression in circulating B-cells, measurement of serum IgG, IgA, and IgM concentration, measurement of antibody responses to vaccination, evaluation of IgG production after cessation of intravenous gamma globulin therapy in patients with clinical indications to discontinue IVIG.
* Evaluate NK cell numbers in long term follow-up of protocol patients. Evaluation will include flow cytometry evaluation of NK cell numbers.
* Determine the vector copy number and the location of vector-integration sites in sorted blood cells. Sorted T-cells, B-cells, NK cells, granulocytes and monocytes will be evaluated for vector copy number. Vector copy number in sorted T-cells will be evaluated as a potential safety measure and will be reported to the FDA if the vector copy number is greater than 5 copies per T cell in any patient at any time. Studies on sorted cells will also include deep sequencing with an automated sequencer to characterize insertion sites, and expression array analysis of T-cell clones to assay for gene expression alterations within 100 kb of the insertion sites.
* Evaluate the overall, long-term safety of lentiviral gene transfer. This will include complete clinical evaluation of any AEs resulting from the gene transfer procedure. If any oncogenic event is seen, this evaluation will include complete molecular characterization of the tumor clone including insertion site analysis, gene expression analysis, and evaluation for the LMO2, Cdkn2a, Notch1, Cyclin D2 gene alterations.

ELIGIBILITY:
Inclusion Criteria:

* Treatment Eligibility Criteria:

* Age <2 years at the time of enrollment.
* No prior therapy with allogeneic stem cell transplantation.
* A clinical diagnosis of SCID-X1 documented in the medical record.
* A proven mutation in the common gamma chain gene as defined by direct sequencing of patient DNA.
* Age > 2 months to < 1 year of age at the time of busulfan administration.
* Less than 300 CD3+ T-cells by flow cytometry or higher if evidence of maternal engraftment as supported by peripheral blood FISH analysis for XY and XX.
* Lymphocyte proliferation to phytohemagglutinin (PHA) <10% of the lower limit of normal for the laboratory.

Treatment Exclusion Criteria:

* Availability of a HLA matched sibling for allogeneic transplantation
* Prior therapy with allogeneic stem cell transplantation
* Positive for HIV infection by genome PCR
* Presence of a medical condition indicating that survival will be less than 16 weeks such as the requirement for mechanical ventilation, severe failure of a major organ system, or evidence of a serious, progressive infection that is refractory to medical therapy.
* The presence of any medical contraindications to general anesthesia and bone marrow harvest by aspiration
* A social situation indicating that the family may not be able to comply with protocol procedures and recommended medical care.

Max Age: 24 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 28 (Estimated)
Dates: Start 2016-08-17 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2034-08 (Estimated)

PRIMARY OUTCOMES:
Number of patients with adequate cell collection and processing | Day 0
  The number of patients who underwent no more than two bone marrow harvests and cryopreservation of at least 1.0 million cells/kg following vector transduction.
Number of patients with adequate neutrophil count recovery after busulfan conditioning | Day 42 post gene transfer
  Adequate recovery is defined as absolute neutrophil count (ANC) >500 cells/μl by day +42 unless the patient is neutropenic prior to busulfan administration.
Number of patients without Grade 4 adverse event (AE) | 42 days post gene transfer
  The number of patients experiencing no directly related grade 4 or greater adverse event.
Number of patients with successful reconstitution | 42 days post gene transfer
  Reconstitution with transduced cells defined as detection of vector-marked peripheral blood cells by real time PCR at or above 0.02% VCN in total WBC.
Number of patients with treatment failure | 42 days post gene transfer
  Treatment failure will be defined as lack of adequate cell collection and processing, lack of neutrophil count recovery by day +42, occurrence of grade 4 or greater toxicities by day +42, and/or lack of detection of >0.02% transduced cells in peripheral blood by day +42 post gene transfer.

OTHER OUTCOMES:
Pharmacokinetic (PK) variables of busulfan | Days -2 and -1 prior to therapy
  Blood collections for pharmacokinetic sampling will be performed with dose 1 and used to determine dose modifications for dose 2, if needed. The specific times for blood collects will be institution specific. Summary statistics will be reported.
Number of patients who achieve the desired therapeutic busulfan AUC | Day 0
  The efficacy of busulfan dose-targeting with busulfan administration every 24 hours for a total of 2 doses in order to achieve a cumulative busulfan AUC of 22 mg*hr/L will be evaluated. The number of patients who achieve the desired therapeutic busulfan AUC will be reported
B-cell function evaluated by Immune response | 52 weeks post gene transfer
  Evaluation may include γc expression in circulating B-cells, measurement of serum IgG, IgA, and IgM concentration, measurement of antibody responses to vaccination, evaluation of IgG production after cessation of intravenous gamma globulin therapy in patients with clinical indications to discontinue IVIG. Summary statistics will be reported.
Number of NK cells | 52 weeks post gene transfer
  Evaluation will include flow cytometry evaluation of NK cell numbers. Summary statistics will be reported.
Vector copy number by location of vector-integration sites in sorted blood cells | up to 10 years post gene transfer
  Sorted T-cells, B-cells, NK cells, granulocytes and monocytes will be evaluated for vector copy number. Studies on sorted cells will also include deep sequencing with an automated sequencer to characterize insertion sites, and expression array analysis of T-cell clones to assay for gene expression alterations within 100 kb of the insertion sites. Summary statistics will be reported.
Event-free survival (EFS) | from baseline up to 10 years post gene transfer
  Event is defined as death, requiring boost post infusion, or an oncogenic event . EFS is defined as time from busulfan infusion to event defined here with all patients surviving at the time of analysis censored.
Overall survival (OS) | up to 10 years post gene transfer
  OS is defined as time from busulfan infusion to death with all patients surviving at the time of analysis censored.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Gottschalk, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (3):
- United States (3):
  - University of California-San Francisco, San Francisco, California
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Seattle Children's Research Institute, Seattle, Washington

REFERENCES:
- [Derived] Mamcarz E, Zhou S, Lockey T, Abdelsamed H, Cross SJ, Kang G, Ma Z, Condori J, Dowdy J, Triplett B, Li C, Maron G, Aldave Becerra JC, Church JA, Dokmeci E, Love JT, da Matta Ain AC, van der Watt H, Tang X, Janssen W, Ryu BY, De Ravin SS, Weiss MJ, Youngblood B, Long-Boyle JR, Gottschalk S, Meagher MM, Malech HL, Puck JM, Cowan MJ, Sorrentino BP. Lentiviral Gene Therapy Combined with Low-Dose Busulfan in Infants with SCID-X1. N Engl J Med. 2019 Apr 18;380(16):1525-1534. doi: 10.1056/NEJMoa1815408. PMID 30995372
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols